CLINICAL TRIAL: NCT01784315
Title: PARASITIC CLEARANCE AND RECURRENCE RATES AMONG PATIENTS WITH VIVAX MALARIA ON CHLOROQUINE AND PRIMAQUINE THERAPY
Brief Title: Parasitic Clearance and Recurrence Rates Among Patients With Vivax Malaria
Acronym: BCAPES
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ministry of Health, Bhutan (Other Government)
Collaborators: Asia Pacific Malaria Elimination Network (Unknown); Menzies School of Health Research (Other)
Responsible Party: Principal Investigator, Dr.Yeshey Dorjey, Principal Investigator, Ministry of Health, Bhutan
Other Study IDs: BCAPES
Record Dates: First submitted 2012-09-01; First posted 2013-02-05 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Parasitemia
Keywords: The presence of parasites in the blood
MeSH Terms: conditions — Parasitemia | interventions — Chloroquine; Primaquine

STUDY DESIGN:
Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — Filter blot paper will be retained to study the whole genome of P.vivax malaria in Bhutan.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chloroquine, primaquine and ACT: Standard dose of Chloroquine( 10mg/kg on day 0 and 5mg/kg on day1 and day2) and Primaquine(0.25mg/kg for 14 days).
  Artemisinin combination therapies (ACT) of 4 tablets on 0,8,24,36,48 and 60 hours will be used for Chloroquine resistant P.vivax infection
  Interventions: Drug: Artemisinin combination therapies (ACT)will be used for Chloroquine resistant P.vivax; Drug: Chloroquine and Primaquine

INTERVENTIONS:
Drug: Artemisinin combination therapies (ACT)will be used for Chloroquine resistant P.vivax — 4 tablets of ACT on 0,8,24,36,48 and 60 hours will be given for Chloroquine resistant P.vivax infection.
  Other Names: ACT
Drug: Chloroquine and Primaquine — Chloroquine:10mg/kg for day1,2 and 5mg/kg for day 3 Primaquine: 0.25mg/kg daily for 14 days.
  Other Names: Chloroquine(CQ); Primaquine (PQ)

SUMMARY:
This research is intended to study the efficacy of CQ alone for P.vivax infection and also to study the recurrence rate among patients with P.vivax on standard dose of CQ and PQ. For this study, PQ will be withheld for 28 days so as to study the efficacy of CQ alone since masking effect over one another was found when CQ is given with PQ. So the investigators are not sure whether the recurrence is due to resistance to CQ or CQ concentration in blood is below therapeutic level or it is due to PQ is in inadequate dose. From this study the investigators will get findings like may be CQ is still working for P.vivax or no longer working for P.vivax due to resistance developed by P.vivax parasites. So for P.vivax which is not responding to CQ therapy, the investigators will go for second line treatment with ACT in a similar fashion as it is given for P. falciparum infection in Bhutan. And if the investigators find CQ is still working for P.vivax infection, the next level of study will be to compare higher dose of PQ with standard dose of PQ ( as practiced now) in lieu of bringing down the relapse rates in P. vivax infection.

DETAILED DESCRIPTION:
In recent time in Bhutan P.vivax infection is on rise compared to other types of malaria like P.falciparum which used to be the most common infections. May be this is mainly due to intensive measures taken place in controlling the diseases especially vector control measures. So that way P.falciparum has gone now. But on other hand P.vivax has peaked the infection. The main reason could be due to resistant to Chloroquine or may be Chloroquine dose is inadequate, and it could also mean it could be due to relapses from the hypnozoites stage where Primaquine dose could be inadequate. Therefore this study is developed to study the efficacy of Chloroquine alone withholding Primaquine for day 28 slightly deviating from the current treatment protocol of Bhutan. That parasitic clearance and recurrence rates will be recorded while on Chloroquine and Primaquine separately. For those patients whose blood stage of parasites doesnt get cleared with standard dose of Chloroquine or for any recurrences occurring before day 28, will be treated with second line treatment with ACT, and the blood level of Chloroquine(drug concentration) will be determined to say whether that could be due to resistance or due to low level of Chloroquine in the blood. And for any recurrences occurring after day 28 while of Primaquine or after completion of Primaquine dosage for a total of 14 days (from day 29 to day 42) those patients will be treated in a similar fashion as initial treatment with Chloroquine and Primaquine and the recurrence rates will be recorded so as to develop next level of study where two different doses of Primaquine (high dose vs low dose) will be compared to study the efficacy of Primaquine.

ELIGIBILITY:
Inclusion Criteria:

* age above 12months
* infection with P.vivax
* presence of axillary temperature >37.5 or history of fever during the past 24h
* ability to swallow oral medication
* ability and willingness to comply with the study protocol for the duration of the study ie 12 months follow up
* informed consent from the patient/parent/guardian in the case of children

Exclusion Criteria:

* signs and symptoms of severe or complicated malaria requiring parenteral treatment according to WHO criteria
* severe malnutrition
* febrile conditions caused by disease other than malaria or other known underlying chronic or severe diseases
* regular medication which interferes with antimalarial pharmacokinetics
* history of hypersensitivity reactions or contraindications to the medicine tested
* positive pregnancy test or breastfeeding
* unable to or unwilling to take contraceptives

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with P.vivax infections from 6 sentinel sites reported to health facility will be recruited for the study after getting the consent signed.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2013-03; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
To measure recurrence rates among patients with vivax malarial infection put on standard dose of Chloroquine and Primaquine | 12 months
  Patients with P.vivax mono-infection will be recruited for the study with a follow up for a period of 12 months. These patients will be put on standard dose of Chloroquine(10mg/Kg on day 0 and 5mg/kg on day 1, and 2) and Primaquine(0.25mg/kg)and any recurrence rates will be measured.

SECONDARY OUTCOMES:
Genotyping of P.vivax strains in Bhutan. | 12 months.
  One time venous blood samples will be collected from patients infected with mixed or mono-infection of P.vivax malaria. And the genotyping will be conducted to study the strains of P.vivax malaria that exist in Bhutan.

OTHER OUTCOMES:
To measure Haemoglobin variations during the malarial infection with treatment. | 12 months.
  Finger prick blood will be taken to check Haemoglobin levels on day 0,3, 7, 14, 28, 35, 42 and at the end of study(ie at the end of 12months).

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Yeshey Dorjey, Principal Investigator — Ministry of Health, Bhutan
Locations (2):
- Bhutan (2):
  - Vector Diseases Control Program, Gelephu, Geylegphug, Gelephu
  - Mr. Thinly, Sarpang, Sarpang District

REFERENCES:
- See also: Related Info — http://www.apmen.org